CLINICAL TRIAL: NCT02826044
Title: Pharmacokinetics,Safety and Tolerability Study Following Single and Multiple Dose of SP2086 in Healthy Volunteers
Brief Title: The Pharmacokinetics Study of Single and Multiple Dose of SP2086 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SP2086-114
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SP2086 50mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 10 healthy volunteers.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086
- SP2086 100mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 10 healthy volunteers.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086
- SP2086 200mg (Experimental): there were 3 groups in the study: 50mg ,100mg and 200mg ,each group including 10 healthy volunteers.All subjects were administrated the medicine at Day 1 and Day 5 to Day 9.During the test,collecting the blood samples were needed before and after taking medicine.
  Interventions: Drug: SP2086

INTERVENTIONS:
Drug: SP2086 — The study has 3 doses groups and the 30 subjects were administrated SP2086 50mg,100mg,200mg respectively.

SUMMARY:
SP2086 is a novel inhibitor of Dipeptide base peptidase 4, allows an insulin-independent approach to improve type 2 diabetes hyperglycemia. In this single-dose and multiple-dose study the investigators evaluated the safety, tolerability and Pharmacokinetics profiles of SP2086 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* BMI(a measure of a person's weight in relation to height)is between 19 and 26 kg/m2,and the weight is equal or less than 100kg.
* without the history of cardiovascular diseases,liver diseases,kidney diseases,gastrointestinal tract diseases,mental nerve diseases and drug allergy.
* Be willing to accept physical contraception.
* Sign the informed consents voluntarily and ensure to completed the study.

Exclusion Criteria:

* Known allergy to SP2086 or any of the excipients of the formulation of SP2086;
* ever occured myocardial infarction,acute coronary syndrome, transient ischemic attack.
* the B hepatitis surface antigen or hepatitis C antibody or syphilis antibody or HIV antibody was positive.
* had participated three or more clinical trial in one year or had participated one time clinical medicine in one month of screening.
* have the history of blood donation in 3 months of screening or received the blood transfusion in 1 months of screening.
* have the history of tobacco,alcohol or drug abuse.
* History of or current clinically significant medical illness as determined by the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of SP2086 | up to Day 13
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086.
The steady-state plasma concentration (Css) of SP2086 | up to Day 13
  Css (a measure of the body's exposure to SP2086) will be compared before and after administration of multiple doses of SP2086
The maximum plasma concentration (Cmax) of SP2086 acid | up to Day 13
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086.
The steady-state plasma concentration (Css) of SP2086 acid | up to Day 13
  Css (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The maximum urine concentration (Cmax) of SP2086 | up to Day 13
  Cmax (a measure of the body's exposure to SP2086) will be compared before and after administration of a single dose of SP2086
The steady-state urine concentration (Css) of SP2086 | up to Day 13
  Css (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
The maximum urine concentration (Cmax) of SP2086 acid | up to Day 13
  Cmax (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of a single dose of SP2086
The steady-state urine concentration (Css) of SP2086 acid | up to Day 13
  Css (a measure of the body's exposure to SP2086 acid) will be compared before and after administration of multiple doses of SP2086
Cumulative excretion of SP2086 | up to Day 13

SECONDARY OUTCOMES:
The number of volunteers with adverse events as a measure of safety and tolerability | up to Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hosital of Jilin University, Changchun, Jilin, China